CLINICAL TRIAL: NCT01718717
Title: Effect of Thoracic Epidural Analgesia for Thoracic Surgery on Arrhythiogenesis
Brief Title: Effect of Thoracic Epidural Analgesia for Thoracotomy on the Occurrence of AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Metaxia Bareka, Anesthesiologist, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TEA and AF
Record Dates: First submitted 2012-10-28; First posted 2012-10-31 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Posterolateral Thoracotomy; Lung Resection; Thoracic Epidural Analgesia; Sympathetic Outflow; Atrial Fibrillation
Keywords: Thoracotomy; Thoracic epidural analgesia; Arrythmiogenesis; Atrial fibrillation; Sympathetic outflow
MeSH Terms: conditions — Atrial Fibrillation | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 6 days TEA (Active Comparator): Postoperative analgesia for the first six postoperative days with TEA and daily monitoring for arrhythmia
  Interventions: Other: Thoracic Epidural Analgesia (TEA)
- 3 days TEA and 3 days intravenous morphine (Active Comparator): Postoperative analgesia for the first three postoperative days with TEA followed for the next three days with intravenous morphine, and daily monitoring for arrhythmia
  Interventions: Other: TEA followed by Intravenous morphine

INTERVENTIONS:
Other: Thoracic Epidural Analgesia (TEA)
  Arms: 6 days TEA
Other: TEA followed by Intravenous morphine
  Arms: 3 days TEA and 3 days intravenous morphine

SUMMARY:
Thoracic epidural anesthesia and analgesia for patients undergoing lung resection can reduce the occurrence of AF if it is continued for six postoperative days instead of just three.

DETAILED DESCRIPTION:
THEA is considered a very effective technique of providing intra and post-operative analgesia for thoracic surgical procedure and it seems that can also be effective in reducing the incidence of postoperative AF in patients undergoing lung resection. Nevertheless the timing of stopping the epidural analgesia and its further substitution with other therapies, remains unclear.

In this study patients who are scheduled for lung resection surgery will undergo the surgery under combined general anesthesia with volatile anesthetics and thoracic epidural anesthesia.

Immediately after surgery the patients will be divided into two groups:

* those who will receive thoracic epidural analgesia for 6 days
* those who will receive thoracic epidural analgesia for 3 days and will then switch to intravenous morphine for another 3 days

All the patients will be monitored daily for arrythmias

ELIGIBILITY:
Inclusion Criteria:

* lung resection
* pneumonectomy

Exclusion Criteria:

* Patient refusal
* AF (present or in the past
* contraindications for epidural catheter placement

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of AF | 6 postoperative days
  Every day, for the first 6 postoperative days, the investigators will record an ECG of the patient, and look after for any presence of AF

SECONDARY OUTCOMES:
Quality of analgesia | 6 postoperative days
  The investigators will record the quality of analgesia, as it can be measured with VAS, for the 6 first postoperative days for all patients

CONTACTS AND LOCATIONS:
Overall Officials: Metaxia Bareka, Medicine, Principal Investigator — Larissa University Hospital; Marina Simaioforidou, Medicine, Study Chair — Larissa University Hospital
Locations (1):
- Larissa University Hospital, Larissa, Thessally, Greece

REFERENCES:
- [Background] Rodgers A, Walker N, Schug S, McKee A, Kehlet H, van Zundert A, Sage D, Futter M, Saville G, Clark T, MacMahon S. Reduction of postoperative mortality and morbidity with epidural or spinal anaesthesia: results from overview of randomised trials. BMJ. 2000 Dec 16;321(7275):1493. doi: 10.1136/bmj.321.7275.1493. PMID 11118174
- [Background] O'Higgins F, Tuckey JP. Thoracic epidural anaesthesia and analgesia: United Kingdom practice. Acta Anaesthesiol Scand. 2000 Oct;44(9):1087-92. doi: 10.1034/j.1399-6576.2000.440909.x. PMID 11028728
- [Background] Mendola C, Ferrante D, Oldani E, Cammarota G, Cecci G, Vaschetto R, Della Corte F. Thoracic epidural analgesia in post-thoracotomy patients: comparison of three different concentrations of levobupivacaine and sufentanil. Br J Anaesth. 2009 Mar;102(3):418-23. doi: 10.1093/bja/aep004. Epub 2009 Feb 3. PMID 19189982
- [Background] De Cosmo G, Aceto P, Gualtieri E, Congedo E. Analgesia in thoracic surgery: review. Minerva Anestesiol. 2009 Jun;75(6):393-400. Epub 2008 Oct 27. PMID 18953284
- [Background] Wildgaard K, Ravn J, Kehlet H. Chronic post-thoracotomy pain: a critical review of pathogenic mechanisms and strategies for prevention. Eur J Cardiothorac Surg. 2009 Jul;36(1):170-80. doi: 10.1016/j.ejcts.2009.02.005. PMID 19307137
- [Background] Scarci M, Joshi A, Attia R. In patients undergoing thoracic surgery is paravertebral block as effective as epidural analgesia for pain management? Interact Cardiovasc Thorac Surg. 2010 Jan;10(1):92-6. doi: 10.1510/icvts.2009.221127. Epub 2009 Oct 23. PMID 19854794
- [Background] Shrivastava V, Nyawo B, Dunning J, Morritt G. Is there a role for prophylaxis against atrial fibrillation for patients undergoing lung surgery? Interact Cardiovasc Thorac Surg. 2004 Dec;3(4):656-62. doi: 10.1016/j.icvts.2004.08.002. PMID 17670334
- [Background] Oka T, Ozawa Y, Ohkubo Y. Thoracic epidural bupivacaine attenuates supraventricular tachyarrhythmias after pulmonary resection. Anesth Analg. 2001 Aug;93(2):253-9, 1st contents page. doi: 10.1097/00000539-200108000-00003. PMID 11473839
- [Background] Simeoforidou M, Vretzakis G, Bareka M, Chantzi E, Flossos A, Giannoukas A, Tsilimingas N. Thoracic epidural analgesia with levobupivacaine for 6 postoperative days attenuates sympathetic activation after thoracic surgery. J Cardiothorac Vasc Anesth. 2011 Oct;25(5):817-23. doi: 10.1053/j.jvca.2010.08.003. Epub 2010 Oct 13. PMID 20947382